CLINICAL TRIAL: NCT04219306
Title: Can a Machine Learning Recognise of Out-of-Hospital Cardiac Arrest During Emergency Calls and Assist Medical Dispatchers
Brief Title: Machine Learning Assisted Recognition of Out-of-Hospital Cardiac Arrest During Emergency Calls.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emergency Medical Services, Capital Region, Denmark (Other Government)
Responsible Party: Principal Investigator, Stig Nikolaj Fasmer Blomberg, PHD-fellow, Emergency Medical Services, Capital Region, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: F-35101-01
Record Dates: First submitted 2019-12-27; First posted 2020-01-07 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Machine learning; Artificial intelligence; Dispatcher assisted telephone CPR; Heart Arrest; Heart Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The study has been designed as a prospective, blinded, randomized clinical trial (RCT). Each call where the machine learning model suspects a cardiac arrest is by lot (1:1) randomized to either alert on dispatchers' screen or no alert on dispatchers' screen
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Machine alert (Experimental): These cardiac suspected cardiac arrest will have had an alert generated by the machine learning model in addition to standard Emergency Medical Services response.
  Interventions: Other: Alert on dispatchers screen 'Suspect cardiac arrest'
- Usual care (No Intervention): These suspected cardiac arrests will receive standard Emergency Medical Services response.

INTERVENTIONS:
Other: Alert on dispatchers screen 'Suspect cardiac arrest' — Alert on dispatchers screen 'Suspect cardiac arrest'
  Arms: Machine alert

SUMMARY:
Emergency medical Services Copenhagen has developed a machine learning model that analyzes the calls to 1-1-2 (9-1-1) in real time. The model are able to recognize calls where a cardiac arrest is suspected. The aim of the study is to investigate the effect of a computer generated alert in calls where cardiac arrest is suspected.

The study will investigate

1. whether a potential increase in recognitions is due to machine alerts or the increased focus of the medical dispatcher on recognizing Out-of-Hospital cardiac Arrest (OHCA) when implementing the machine
2. if a machine learning model based on neural networks, when alerting medical dispatchers will increase overall recognition of OHCA and increase dispatch of citizen responders.
3. increased use of automated external defibrillators (AED), cardiopulmonary resuscitation (CPR) or dispatch of citizen responders in cases of OHCA on machine recognised OHCA vs. medical dispatcher recognised OHCA.

DETAILED DESCRIPTION:
Chances of survival after out-of-hospital cardiac arrest decrease 10% per minute from collapse until CPR is initiated. dispatcher assisted telephone CPR will be initiated only in cases where the dispatcher recognizes the cardiac arrest.

In a previous project "Can a computer through machine learning recognise of Out-of-Hospital Cardiac Arrest during emergency calls" (supported by TrygFoundation), the investigators found, it was possible to create a Machine Learning (ML) model, which could recognise OHCA with higher precision than medical dispatchers at the Emergency Medical Dispatch Center (EMDC-Copenhagen).

In this study the model andt is effect is to be documented in the EMDC-Copenhagen. For this purpose, a computer server running the ML-model are created. This server is integrated in the network at EMDC-Copenhagen, making it possible to push alerts to the medical dispatcher, when a cardiac arrest is recognised by the model.

With aid of machine learning, the hypothesis is, that recognition of OHCA is improved, and happen both more frequent and faster than present.

An instruction for the medical dispatchers is developed, which guides the medical dispatcher in instance of an alert from the machine.

ELIGIBILITY:
Inclusion Criteria:

* Call regarding a cardiac arrest registered in the national Danish Cardiac Arrest Registry
* OHCA is recognized by machine-learning model
* Call originates from 1-1-2

Exclusion Criteria:

* OHCA Emergency Medical Services - witnessed
* Call is from another authority (police or fire brigade)
* Call is a repeat call
* Call has been on hold for conference

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5242 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Dispatcher recognition of cardiac arrest | During call to emergency Medical Services, up to 15 minutes from call start.
  Dispatcher recognition of out-of-hospital cardiac arrest is the primary outcome. Recognition is reported by a questionnaire filled in by a group of auditors listening to recordings of all included calls. The questionnaire is a modified CARES protocol for the calls and consists of 21 questions whereby the quality of the call is evaluated. The questionnaire is validated and has been used in other studies.

SECONDARY OUTCOMES:
Time to recognition | During call to emergency Medical Services, up to 15 minutes from call start.
  Time from call-start until dispatcher recognition of cardiac arrest
Dispatcher assisted telephone CPR | During call to emergency Medical Services, up to 15 minutes from call start.
  Does the dispatcher ask caller to initiate CPR.
Time to T-CPR | During call to emergency Medical Services, up to 15 minutes from call start.
  Time from call-start until dispatcher starts guiding caller in cpr

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Lippert, MD, Study Director — Copenhagen Emergency Medical Services
Locations (1):
- Emergency Medical Services Copenhagen, Ballerup Municipality, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Data will be available upon reasonable request by mail to primary investigator.

REFERENCES:
- [Background] Blomberg SN, Folke F, Ersboll AK, Christensen HC, Torp-Pedersen C, Sayre MR, Counts CR, Lippert FK. Machine learning as a supportive tool to recognize cardiac arrest in emergency calls. Resuscitation. 2019 May;138:322-329. doi: 10.1016/j.resuscitation.2019.01.015. Epub 2019 Jan 18. PMID 30664917
- [Derived] Blomberg SN, Christensen HC, Lippert F, Ersboll AK, Torp-Petersen C, Sayre MR, Kudenchuk PJ, Folke F. Effect of Machine Learning on Dispatcher Recognition of Out-of-Hospital Cardiac Arrest During Calls to Emergency Medical Services: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jan 4;4(1):e2032320. doi: 10.1001/jamanetworkopen.2020.32320. PMID 33404620

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT04219306/Prot_SAP_000.pdf